CLINICAL TRIAL: NCT06332183
Title: Genome-wide Association Study (GWAS) and Epigenome-wide Association Study (EWAS) in Patients With Erdheim-Chester Disease
Brief Title: GWAS and EWAS in Patients With Erdheim-Chester Disease
Status: Recruiting | Type: Observational
Sponsor: Augusto Vaglio (Other)
Responsible Party: Sponsor-Investigator, Augusto Vaglio, Associate Professor of Nephrology, Principal Investigator, Meyer Children's Hospital IRCCS
Organization: Meyer Children's Hospital IRCCS (Other)
Other Study IDs: ECDGWAS
Record Dates: First submitted 2024-02-21; First posted 2024-03-27 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Erdheim-Chester Disease
MeSH Terms: conditions — Erdheim-Chester Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Presence of polymorphisms: Statistical analysis of GWAS data, Genome-wide methylation pattern analysis, Integration of GWAS data and methylation data (meQTL analysis), Pathway enrichment analysis
  Interventions: Genetic: Presence of polymorphisms

INTERVENTIONS:
Genetic: Presence of polymorphisms — Statistical analysis of GWAS data, Genome-wide methylation pattern analysis, Integration of GWAS data and methylation data (meQTL analysis), Pathway enrichment analysis

SUMMARY:
Erdheim-Chester Disease (ECD) is a rare form of histiocytosis characterized by the proliferation of blood cells, known as histiocytes, which infiltrate various organs and tissues, often causing irreversible damage. The causes of the condition are still unknown, and although some mutations in genes involved in cell proliferation have been identified, other factors may be involved. Susceptibility to developing rare diseases like ECD is typically associated with genetic factors, including DNA polymorphisms and epigenetic modifications.

This study aims to analyze the entire genome of a large cohort of patients with ECD and healthy controls to determine whether there are polymorphisms and epigenetic variants associated with susceptibility to developing the disease. The study could thus clarify the genetic predisposition to ECD development, provide insights into disease pathogenic mechanisms, and identify proteins or cellular mechanisms potentially targeted by specific treatments.

ELIGIBILITY:
Inclusion Criteria:

- ECD with histological confirmation of disease

Exclusion criteria:

- previously treated patients (for methylation and gene expression)

Ages: 1 Year to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Incident and prevalent patients with ECD
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2019-07-17 (Actual); Primary Completion 2024-07-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
Polymorphisms and genetic variants correlated with disease development | 5 years
  To investigate the presence of polymorphisms and genetic variants correlated with disease development, through a GWAS study. This task will be carried out by analyzing the frequency of the identified polymorphisms in patients and controls
Methylation in Erdheim-Chester disease | 5 years
  To identify differences in gene methylation between patients with ECD and healthy controls, through an EWAS study. This task will be carried out by analyzing the grade of methylation in patients and controls
Gene expression in Erdheim-Chester disease | 5 years
  To investigate the correlation between genetic variants or epigenetic profiles associated with the disease (previous outcomes) and specific clinical manifestations (organ involvement, somatic mutations, response to treatment, survival)

CONTACTS AND LOCATIONS:
Locations (5):
- Hopital Pitié Salpetrière, Paris, France
- Italy (3):
  - Meyer Children's Hospital IRCCS, Florence
  - IRCCS Ospedale San Raffaele, Milan
  - AOU Parma, Parma
- Genetics Lab, CSIC, Granada, Spain

IPD SHARING:
Plan to Share IPD: No